CLINICAL TRIAL: NCT00216801
Title: The Relationship of Ochratoxin A to Upper Tract TCC Malignancies, Testicular Cancer, and Renal Cell Cancer
Brief Title: Relationship of Ochratoxin A to Upper Urologic Cancers
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Dr. S. Pautler, Lawson Health Research Institute
Other Study IDs: R-05-082; 11293
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Transitional Cell Carcinoma; Renal Cell Cancer; Testicular Cancer
Keywords: Upper Tract Transitional Cell (TCC)
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This pilot study will explore the relationship of Ochratoxin A (OTA) levels in patients with upper tract transitional cell (TCC), renal cell, and testicular cancers by measuring levels of OTA in serum and tumor samples. Dietary exposure will also be analyzed.

DETAILED DESCRIPTION:
Ochratoxin A (OTA, a ubiquitous mycotoxin) is a common food contaminant that enters the food chain from plants such as cereals. OTA can be inhaled or ingested and livestock and humans feeding on OTA contaminated food have been found to have detectable levels of this chemical in their sera, liver, and kidneys.

There is risk for occupational and environmental exposure to OTA. Thus, exposure to this mycotoxin may be a poorly recognized problem in our society. OTA has been classified as a group 2b possible carcinogen. Exposure to OTA has been implicated in teratogenesis (fetal malformation), nephrotoxicity, gonadotoxicity and carcinogenesis. The mechanisms for these effects of OTA have not been fully explained. There is an increasing incidence of testis cancer in Western societies combined with the increasing OTA exposures being reported. As well as studying the relationship of OTA to TCC initially, we also plan to examine a possible relationship between OTA and testicular cancer as well as renal cell carcinoma (RCC). To date, very little research into the effects of mycotoxins in humans has been performed. We plan to apply proven techniques of serum analysis using:

1. ELISA or Enzyme Linked Immuno-absorbent Assay which is used to measure the presence of an antibody or antigen in the bloodstream
2. Immunohistochemistry (pathological analysis from resected tumors)
3. High -pressure liquid chromatography (HPLC) of tumor tissue to investigate the role of OTA in human genitourinary cancers. A group of subjects without cancer will be used as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Study Group

  1. Informed consent
  2. Must have resectable non-metastatic upper tract transitional cell carcinoma, renal cell carcinoma, or testicular carcinoma.
  3. Willingness to be followed for survival data.
* Control Group

  1. Informed consent
  2. No history of carcinoma

Exclusion Criteria:

1. Metastatic upper tract transitional cell carcinoma, renal cell carcinoma, or testicular carcinoma.
2. Any other ongoing or previous malignancy other than basal or squamous cell skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Must have resectable non-metastatic upper tract transitional cell carcinoma, renal cell carcinoma, or testicular carcinoma.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pautler, MD, FRCSC, Study Director — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St. Josephs Health Care, London, Ontario, Canada